CLINICAL TRIAL: NCT03605511
Title: A Observational Study to Determine the Prevalence of Pregnancy-related Thrombotic Thrombocytopenic Purpura and Atypical Haemolytic Uraemic Syndrome in Women Affected by Specific Obstetric Complications
Brief Title: TTP and aHUS in Complicated Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0217
Record Dates: First submitted 2018-07-02; First posted 2018-07-30 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-07

CONDITIONS: Thrombotic Thrombocytopenic Purpura; Atypical Hemolytic Uremic Syndrome; Pre-Eclampsia; HELLP Syndrome; Thrombocytopenia; IUGR; Stillbirth; Thrombotic Microangiopathies
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic; Atypical Hemolytic Uremic Syndrome; Pre-Eclampsia; HELLP Syndrome; Thrombocytopenia; Stillbirth; Thrombotic Microangiopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ADAMTS 13, complement and angiogenic biomarkers — ADAMTS 13, complement and angiogenic biomarkers

SUMMARY:
A single site observational study aiming to:

(i) Identify cases of previously undiagnosed thrombotic thrombocytopenic purpura (TTP) and atypical haemolytic syndrome (aHUS) in a cohort of women with complicated pregnancies (ii) Characterise the clinical features of these cases and (ii) Identify clinical features or biomarkers which may help distinguish TTP/aHUS from other complications of pregnancy such as preeclampsia

ELIGIBILITY:
Inclusion Criteria:

- Women, either currently pregnant or recently postpartum, and affected by one or more of the following complications in the index pregnancy: (i) Preeclampsia with evidence of end organ damage (renal/ liver/ haematological/ neurological) or uteroplacental dysfunction (FGR/IUFD) (ii) HELLP syndrome (iii) Fetal growth restriction (FGR) (growth <10th centile) that is unexplained (ie not due to infection, fetal structural anomaly, fetal chromosomal or pre-existing maternal medical problem) (iv) Intrauterine fetal demise (IUFD) after 20 weeks' gestation that is unexplained (v) Unexplained new onset renal impairment (defined by serum creatinine >85umol/L 1st trimester, or >80umol/L 2nd trimester, or >90 umol/L 3rd trimester[32]; OR an increase in serum creatinine by (i) at least 1.5 times the baseline or (ii) of equal or greater than 26.5umol/L (as per KDIGO criteria) (vi) Unexplained new onset thrombocytopenia (platelets <75x10^9/L)

Exclusion Criteria:

* Previous diagnosis of TTP or aHUS
* Known disorder of complement dysregulation
* Patients not wishing to participate
* Patients aged less than 16
* Patients lacking capacity to provide informed consent

Min Age: 16 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All women receiving obstetric care at University College Hospitals London NHS Trust over the study period
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-03-14 (Estimated); Study Completion 2020-03-14 (Estimated)

PRIMARY OUTCOMES:
Frequency of TTP and aHUS in the cohort | At study completion, approximately 18 months after recruitment of first patient
  Number of new cases identified as a percentage of sample size

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom